CLINICAL TRIAL: NCT04821869
Title: ProAir Digihaler in COPD Disease Management: A Real World Study to Assess ProAir Digihaler Inhalation Parameters Thresholds and Their Use to Identify Deterioration in Clinical Practice
Brief Title: ProAir Digihaler in COPD Disease Management: A Real World Study
Status: Completed | Type: Observational
Sponsor: Pulmonary Research Institute of Southeast Michigan (Other)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 002
Record Dates: First submitted 2021-03-19; First posted 2021-03-30 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2022-04

CONDITIONS: COPD; COPD Exacerbation Acute
Keywords: COPD; Digihaler; Rescue Medication; Disease Management
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Drug: ProAir Digihaler — Monitor parameters transmitted from the Proair Digihaler to the Digihaler Dashboard, including peak inspiratory Flow, inspiratory volume and frequency of rescue use
  Other Names: Digihaler Device
Device: Digihaler — Monitor parameters transmitted from the Proair Digihaler to the Digihaler Dashboard, including peak inspiratory Flow, inspiratory volume and frequency of rescue use
  Other Names: Digihaler Dashboard

SUMMARY:
A pilot study to explore the utilization of the TEVA ProAir Digihaler rescue medication use and inhalation parameters to identify disease deterioration to help in the management of COPD patients in clinical practice. The study is designed to follow a small sample size of patients with COPD, monitor and collect inhalation parameters from the Digihaler dashboard, and changes in symptom control as measured by the COPD Assessment Test (CAT) to identify potential inhalation parameter thresholds that could be applied to the management of patients with COPD in clinical practice.

DETAILED DESCRIPTION:
The trial is an unblinded open label single center study designed to identify trends in Peak Inspiratory Flow (PIF) rates and Rescue Albuterol Inhaler usage (Inhalations) that associate with disease deterioration as defined by worsening of symptoms and reduced lung function in patients with COPD.

The study will consist of a run-in period of approximately 2 weeks, a treatment period of 6 months and a follow-up period of 1 week. Twenty (20) patients with COPD requiring intermittent short acting beta agonist (SABA) rescue inhaler usage, but not requiring frequent SABA nebulizer rescue usage, will be enrolled.

After signing informed consent, patients will undergo a screening evaluation. During the run-in period, patients will continue on their COPD maintenance treatments, while discontinuing all previously prescribed periodic use rescue medications. Upon completion of screening, all patients will be dispensed a ProAir Digihaler to be used exclusively as their rescue medication throughout the duration of the study. During the run-in period all rescue inhaler usage will be electronically monitored and patient data from the Digihaler Dashboard will be downloaded every other business day basis (Monday, Wednesday and Friday).

At the completion of at least 2 weeks of run-in (with a minimum of at least 8 rescue inhaler usages) and with documentation of stable clinical status throughout run-in, the patient will return for baseline testing; including vital signs, health related quality of life and Anthonisen Exacerbation questionnaires, pre and post bronchodilator spirometry and 6-minute walk testing (see table/flow chart). Average Peak Inspiratory Flow (Baseline PIF) and average Number of Rescue Inhalations per day (Baseline Inhalations) will be determined from the Digihaler Dashboard Data downloads during run-in.

In the event that the patient does not meet number of rescue inhaler usages or does not have a stable clinical status during run-in, an additional 2 weeks of run-in may be obtained. If at the end of the extended run-in period so that Baseline PIF and Baseline Inhalations cannot be determined or the patient continues to be clinically unstable, the patient will be discontinued from the study. If the patient has an upper respiratory tract infection or COPD exacerbation during run-in, they will also be discontinued from the study. Patients may be re-screened one time at a later date, when stable.

Once run-in and baseline testing are complete, all patients will continue on their maintenance COPD medications and use the ProAir Digihaler rescue SABA exclusively for the next 6 months. Patients will be provided with paper forms of the CAT, BCSS and Anthonisen Exacerbation criteria, to be completed at home on a weekly basis and mailed to the research center upon completion).

Throughout the treatment period, all rescue inhaler usage will be electronically transmitted to, monitored at and downloaded from the Digihaler Dashboard by the research center on every other business day basis (Monday, Wednesday and Friday). At the completion of each Digihaler Dashboard Data Download, comparisons of Daily PIF (average PIF of all rescue inhalations in a day) and Daily Inhalations (number of rescue inhalations in a day) to Baseline PIF and Baseline Inhalations will be made.

All patients with Daily Inhalations exceeding Baseline Inhalations by ≥4 Inhalations per day and/or with a Daily PIF ≤80% of Baseline PIF for 2 consecutive days will be DEFINED as "at risk". For each "at risk" event, the patient will be contacted, their health status reviewed, and CAT and Anthonisen Exacerbation questionnaires will be administered. Based on symptoms, patients may also be advised to seek additional medical care.

All patients will be contacted on a monthly basis, irrespective of "risk" findings and seen in person every 3 months. All medication usage (including ProAir Digihaler medication usage), changes in medical care, healthcare contacts and usage, and any adverse events will be recorded. All office records for the intervening time period will be reviewed and Information for any non-office healthcare contacts and usage will be requested to provide detailed clinical information for comparison to Digihaler usage records.

At months 3 and 6 on treatment, all subjects will return to the research center, where vital signs, Anthonisen Exacerbation and CAT questionnaires, and post bronchodilator spirometry will be assessed. All medication usage (including ProAir Digihaler medication usage), changes in medical care, healthcare contacts and usage, and any adverse events will be recorded. All office records for the intervening time period will be reviewed and Information for any non-office healthcare contacts and usage will be requested to provide detailed clinical information for comparison to Digihaler usage records. Three (3) new ProAir Digihalers will be dispensed at month 3.

Throughout the treatment period, all rescue inhaler usage will be electronically monitored and downloaded from the Digihaler Dashboard by the research center on an every other business day basis (Monday, Wednesday and Friday). At the completion of each Digihaler Dashboard Data Download, comparisons of Daily PIF (average PIF of all rescue inhalations in a day) and Daily Inhalations (number of rescue inhalations in a day) to Baseline PIF and Baseline Inhalations will be made.

All patients with Daily Inhalations exceeding Baseline Inhalations by ≥4 Inhalations per day and/or with a Daily PIF ≤80% of Baseline PIF for 2 consecutive days will be DEFINED as "at risk". For each "at risk" event, the patient will be contacted, their health status reviewed, and CAT and Anthonisen Exacerbation questionnaires will be administered. Based on symptoms, patients may also be advised to seek additional medical care.

At the conclusion of the 6-month treatment period the patients will return to the research center for a final visit, returning all study medication not previously returned. The patient will be advised to resume usage of their prior rescue inhaler medication at that time. A telephone call will be made to the patient 1 week after their final in-person visit, to assess vital status and any adverse events that may have occurred subsequent to discontinuing the ProAir Digihaler.

ELIGIBILITY:
Inclusion Criteria:

1. Documented history of COPD by ATS/GOLD criteria
2. Age > 45 years
3. Patient willing and able to:

   1. participate in the study, including all scheduled visits
   2. demonstrate the ability to use the ProAir Digihaler, including transfer of Digihaler data via blue-tooth to a smart device
   3. perform all required testing, including spirometry and walk tests
   4. complete all home questionnaires and participate in all telephone contacts
   5. switch current rescue inhaler/device to ProAir Digihaler
4. Baseline spirometry consistent with COPD (post bronchodilator FEV1 < 80% predicted, FEV1/FVC <70%)
5. Use of albuterol inhaler as primary device for administration of rescue therapy
6. Reported use of rescue inhaler at least twice (4 inhalations) a week in the previous 6 months
7. Access to smartphone with blue-tooth and cellular/internet access

Exclusion Criteria:

1. Allergy, contraindication or inability to use albuterol sulfate
2. Frequent use of a nebulizer as rescue therapy (>1 time per day)
3. Current diagnosis of asthma
4. Unstable medical condition that could prevent the completion of the research trial
5. Pregnancy, planning to become pregnant or breast feeding
6. Failure to use rescue inhaler during Run-in period (minimum of at least 8 rescue inhaler inhalations over the 2 weeks)
7. Exacerbations that require discontinuation from study (during run-in period)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with COPD
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary T Ferguson, M.D., Principal Investigator — Pulmonary Research Institute of Southeast Michigan
Locations (1):
- Pulmonary Research Institute of Southeast Michigan, Farmington Hills, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Data limited to study collaborative research organizations only

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment initiated May 19, 2021. Study completed June 20, 2022. The study was conducted at a single clinical research center, the Pulmonary Research Institute of Southeast Michigan.
Pre-assignment Details: 27 subjects were recruited and consented to enroll 20 subjects for 6 months of observation. 7 participants failed during run-in: 4 due to COPD exacerbation during run-in, 1 did not meet FEV1 entry criteria and 2 withdrew during run-in unrelated to study participation. All 20 participants enrolled in the study completed the study and were included in all analysis.Post study, subjects were stratified based on the occurrence of a COPD exacerbation during the study and analyzed accordingly.
Groups:
- Digihaler Device User: Single arm pilot study assessing the relationship of deterioration in COPD healthcare status (COPD exacerbations and/or worsening in COPD Assessment Test ≥2) to changes in physiologic parameters measured from usage of an albuterol Digihaler inhalation device, including peak inspiratory flow (PIF), extra inhaler puff usage per day and inhalation volume (InV) prior to any heaalthcare deterioration event.
Period: Overall Study
Arm/Group | Digihaler Device User
Started | 27
Post run-in Enrollment (Met all inclusion/exclusion criteria post run-in) | 20
Completed | 20
Not Completed | 7
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 2
Not completed — Did not meet FEV1 criteria | 1

BASELINE CHARACTERISTICS:
Population: All subjects meeting inclusion/exclusion criteria
Groups:
- Subjects With COPD Exacerbations: All subjects meeting inclusion exclusion criteria who had an exacerbation during the study
- Subjects With no COPD Exacerbation: All subjects meeting inclusion exclusion criteria who did not have an exacerbation during the study
- Total: Total of all reporting groups
Arm/Group | Subjects With COPD Exacerbations | Subjects With no COPD Exacerbation | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 5 | 4 | 9
Age, Continuous [Mean (Full Range); unit: years] | 66 [57 to 74] | 67 [57 to 78] | 67 [57 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 2 | 6 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20
Baseline PIF [Mean (Standard Deviation); unit: L/min] — Peak Inspiratory Flow (PIF) is the maximal inspiratory flow a subject is able to generate while inspiring through a dry powder inhaler (or other inspiratory flow measurement tool)
  L/min | 73.6 (23.2) | 66.2 (18.3) | 70.3 (21.0)

OUTCOME MEASURES:

1. Primary Outcome: PIF Alerts and COPD Exacerbations
Description: Presence of a Peak Inspiratory Flow (PIF) alert prior to a COPD Exacerbation
  Peak Inspiratory Flow (PIF) is the maximal inspiratory flow achieved during each patient inhalation of the Digihaler dry powder inhaler. PIF is automatically measured by the Digihaler dry powder inhaler during every inspiration of medication by a subject. Inspiratory flow is used to inhale respiratory medications into the lungs. A low inspiratory flow rate has been considered to place a COPD patient at risk for reducing medication inhalation and for other adverse outcomes. An acute fall in a patient's PIF may also be a marker of an impending change in a patient's condition.
  All acute COPD exacerbations were assessed by patient history, diaries and direct patient interviews. If a COPD Exacerbation had occurred, PIF measurements in the prior 2 weeks were assessed to determine if a PIF Alert, defined as a 20% fall in PIF from baseline for a minimum of 2 consecutive days, had occurred in the 2 weeks prior.
Time Frame: 6 months
Population: This was an observational study with one treatment arm using a single study drug during the 6 months of study. All acute COPD exacerbation events meeting Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria for an acute COPD exacerbation were assessed to determine if a PIF alert was present prior to the event. All subjects/ events were assessed as a treatment outcome (not a treatment arm).
Measure: Number; unit: Low PIF Alert
Units Other Than Participants: COPD Exacerbations
Groups:
- COPD Exacerbation: All events meeting GOLD criteria for an acute COPD exacerbation
Arm/Group | COPD Exacerbation
Number analyzed (Participants) | 20
Number analyzed (COPD Exacerbations) | 22
Low PIF Alert | 2

2. Primary Outcome: Low PIF Alerts and Worsening CAT Score
Description: Presence of a Low Peak Inspiratory Flow (PIF) alert, defined by an 20% reduction in PIF from baseline for a minimum of 2 consecutive days occurring in the 2 weeks prior to a worsening of a subject COPD Assessment Test Score (CAT, score range 0-40, clinically important difference defined as a change in CAT score of 2 or more over time with an increase in value identifying worsening disease).
  Peak Inspiratory Flow (PIF) is the maximal inspiratory flow achieved during each patient inhalation of the Digihaler dry powder inhaler. PIF is automatically measured and recorded by the Digihaler device during every inspiration of medication with the device. All PIF measures in the 2 weeks prior to any worsening of CAT were assessed and a PIF alert was identified as being present if PIF fell by ≥20% from baseline on 2 or more consecutive days in the 2 weeks prior to a worsening of CAT score event.
Time Frame: 6 months
Population: All worsening of CAT score events
Measure: Number; unit: Low PIF Alert
Units Other Than Participants: Worsening of CAT
Groups:
- Worsening CAT Score: All events identified as a Worsening of CAT score ≥2 unit event
Arm/Group | Worsening CAT Score
Number analyzed (Participants) | 20
Number analyzed (Worsening of CAT) | 40
Low PIF Alert | 3

3. Secondary Outcome: Rescue SABA Puff Use Alerts and COPD Exacerbations
Description: Presence of a Rescue SABA Puff Use Alert, defined as an increase of 2 or more rescue inhaler puffs per day above baseline for 2 or more days in the 2 weeks prior to any COPD exacerbation. Rescue SABA Puff use is the counted and recorded use of the DIgihaler inhaler device each time the subject uses of the Digihaler device.
Time Frame: 6 months
Population: All acute COPD exacerbation events meeting Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria for an acute COPD exacerbation.
Measure: Number; unit: Rescue SABA Puff Use Alert
Units Other Than Participants: COPD Exacaerabations
Arm/Group | COPD Exacerbation
Number analyzed (Participants) | 20
Number analyzed (COPD Exacaerabations) | 22
Rescue SABA Puff Use Alert | 0

4. Secondary Outcome: Low IV Alerts and COPD Exacerbations
Description: Presence of a Low Inhalation Volume (IV) alert, defined by a 20% fall in IV from baseline for 2 or more days in the 2 weeks prior to any COPD exacerbation. IV is the volume of air inhaled and measured during each patient inhalation use of the Digihaler device.
Time Frame: 6 months
Population: as for outcome 3
Measure: Number; unit: Low IV Alert
Units Other Than Participants: COPD exacerbation
Arm/Group | COPD Exacerbation
Number analyzed (Participants) | 20
Number analyzed (COPD exacerbation) | 22
Low IV Alert | 4

ADVERSE EVENTS:
Time Frame: Data was collected from consent to post study follow-up over approximately 7 months
Description: All ad verse event descriptions and definitions are per clinicaltrials.gov
Arm/Group | Digihaler Device User
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 3/27
Other Adverse Events (participants affected / at risk) | 16/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digihaler Device User (N=27)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 (4) — Worsening of COPD requiring hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digihaler Device User (N=27)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 12 (18) — COPD exacerbation requiring medical intervention
Non respiratory adverse events (General disorders) | 12 (12) — Any ev ent qualifying as an adverse event that was not a COPD exacerbation AE

LIMITATIONS AND CAVEATS:
This study was not designed for or intended to evaluate the use of the Digihaler to predict future clinical events in COPD patients. Rather, it was a non-powered exploratory pilot study designed to provide preliminary information and insights that might serve as the basis for future studies to assess whether the use of rescue albuterol in a digital inhaler device could be used as a predictive tool.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT04821869/Prot_000.pdf
  • Informed Consent Form (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT04821869/ICF_001.pdf